CLINICAL TRIAL: NCT05646875
Title: A Comprehensive Evaluation of Hyperbaric Oxygen Therapy in Resuscitation Medicine - a Pilot Study (HOT-RESUS 1 Trial)
Acronym: HOT-RESUS 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Koen Monsieurs, Prof. Koen Monsieurs, MD, University Hospital, Antwerp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HOT-RESUS 1
Record Dates: First submitted 2022-11-22; First posted 2022-12-12 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Heart Arrest; Brain Injuries
MeSH Terms: conditions — Heart Arrest; Brain Injuries | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: 3 groups: 1) post-ROSC patients 2) cardiac arrest survivors already discharged 3) healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- post-ROSC (Experimental): patients directly post-ROSC receiving HBOT
  Interventions: Other: hyperbaric oxygen therapy
- cardiac arrest survivors discharged home receiving HBOT (Active Comparator): cardiac arrest survivors discharged home
  Interventions: Other: hyperbaric oxygen therapy
- healthy volunteers receiving HBOT (Active Comparator): healthy volunteers receiving HBOT
  Interventions: Other: hyperbaric oxygen therapy

INTERVENTIONS:
Other: hyperbaric oxygen therapy — Hyperbaric oxygen therapy in a pressurized chamber, duration 1-2 hours at 2-3 ATA

SUMMARY:
In this prospective pilot study, the effects of hyperbaric oxygen therapy (HBOT) in post-cardiac arrest syndrome will be evaluated. However, the primary outcome of this pilot study will be the feasibility of this approach. If feasibility is determined, a larger study with adequate powering is to follow.

DETAILED DESCRIPTION:
Cardiac arrest (CA) necessitating cardiopulmonary resuscitation (CPR) currently results in a survival rate of around 8% in Europe. The much lower percentage of patients being discharged from hospital with a favourable neurological outcome or with a satisfactory degree of quality of daily life still shows room for improvement in post CA care. The so- called post-CA syndrome after return of spontaneous circulation (ROSC) requires a multidisciplinary management in a coordinated fashion. Despite steady advances in this very specific field of intensive care medicine, both neurologic and psychologic disability after CA still remain dismal with hypoxic brain injury as the main determinant (primary cause of death in 68 % of in-hospital CA and 23 % of out-of-hospital CA [OHCA]), and the optimal treatment approach might still be missing additional beneficial therapeutic options. The neuropathology of anoxic brain injury includes neural toxicity, intracellular calcium accumulation, oxygen free radicals, excitatory amino acid release, reperfusion injury and endothelial dysfunction, with a clinical presentation through impairment of visual, perceptive, expressive, cognitive, and motor functions, or psychological distress. As voiced by former patients and relatives, those functional outcomes are of utmost importance. Therefore, the Core Outcome Set for Cardiac Arrest (COSCA) was developed.

Hyperoxia vs. hyperbaric oxygenation therapy: It seems intuitive that a hypoxic or anoxic state such as CA necessitates a hyperoxic environment for convalescence. However, hyperoxia has been proven to be harmful, mostly through systemically accumulating reactive oxygen species (ROS), inducing oxidative stress in cellular structures, contributing to deleterious cell dysfunction and apoptosis induction, and finally leading to unfavourable neurological outcomes. Hyperoxia is advised against in current guidelines, but not defined or described in detail, leaving clinicians without a clear recommendation. In parallel, hyperbaric oxygen therapy (HBOT) was in its beginnings thought to facilitate similar effects. However, HBOT was then slowly researched in more detail, leading to a paradoxon: On the one side, the described harmful effects of hyperoxia are known, on the other side HBOT was shown to provide antioxidant effects, balancing out the negative features. HBOT has thus been described as safe due to its balance between oxidation and antioxidation. Key molecular changes following HBOT include a preservation of mitochondrial properties (e.g., through upregulation of ATP production), a reduction of neuroinflammatory processes (e.g., through reduced cytokine secretion), an upregulation of angiogenesis (e.g., through an upregulation of cerebral blood flow and vascular endothelial growth factor [VEGF], or downregulation of metalloproteinases), suppression of neutrophil-endothelial adhesion, and the mentioned upregulation of both ROS and antioxidants. HBOT has been shown to restore and increase perfusion and oxygenation of at-risk tissue, to enhance cerebral microcirculation and stabilize the blood-brain barrier through metalloprotease regulation, and to decrease intracranial pressure and cerebral edema. Moreover, it has been linked to several pathways leading to a preservation of neural tissue and a reduction of apoptosis, for instance shown via reduced levels of hypoxia-inducable factor 1 alpha (HIF1α). HBOT has also been linked to anti-inflammatory effects, for instance through a decrease in tumor necrosis factor alpha (TNFα) or an inhibition of the accumulation of leukocytes in ischemic areas. Mentionable other beneficial results of HBOT include improvement of left ventricular function, or the induction of significant senolytic effects including increasing telomere length and clearance of senescent cells. HBOT has in the past been used quite successfully in animal and human ischemic stroke patients for stimulation of a hyperoxic environment during ischemic and reperfusion periods, for instance leading to a reduced infarction area and neuronal death reduction. It was even demonstrated that cognitive function could be improved, and it was hypothesized that it could signal-induce the (re-)growth of grey and white cerebral matter. Moreover, HBOT might have the potential to re-gain suppressed psychological properties such as memories through a complex mechanism of increased cerebral tissue oxygenation, or even to induce an enhanced multitasking performance in healthy volunteers. A recent review on the impact of HBOT on cognitive functions yielded controversial results, concluding with a call for more standardized outcome evaluation.

So far, only four studies and one case report assessed HBOT around CA: In 1952, Koch et al. described a case of CA and cerebral edema being treated with HBOT "successfully". However, the given information lacks detail and is highly out-dated. In 1982, Kapp et al. subjected cats to CA and HBOT, observing a beneficial modification of functional impairment and metabolic derangements. Rosenthal et al. showed in 2003 that HBOT could inhibit neuronal death and improve neurologic outcomes after CPR in a canine model, concluding that HBOT has the potential of overcoming postresuscitative delivery-dependent cerebral ischemia. Of utmost importance, the authors could demonstrate that only one exposure to hyperbaric conditions was sufficient to show an effect, and they proved that HBOT is also beneficial in a globally ischemic model as opposed to a vessel-occluded model such as in the majority of studies covering stroke patients. Van Meter et al. assessed HBOT during CA (and ongoing cardiopulmonary resuscitation) in a porcine model, and concluded that the rate of sustained ROSC was higher in a high-dose HBOT regimen than in a low-dose one or in controls. The same authors even hypothesized HBOT to be potentially feasible for a more widespread use in CA patients in the future. Hadanny et al. investigated eleven human CA survivors receiving HBOT in 2015, and found that the treatment significantly improved memory, attention and executive functions evaluated via NeuroTrax®, a validated psychologic test series. The findings correlated with increased activities in the respective brain areas in imaging. Further research was recommended, but never conducted. Apart from these data, cases on HBOT after CA due to carbon monoxide poisoning exist, but focus on the treatment of this intoxication per se and not on other effects. Interestingly, HBOT was also shown to be stimulating the regeneration of peripheral nerval function after brain injury, potentially inhibiting the development of polyneuropathy and/or improving motor function after CA.

Assessing HBOT effects: In terms of assessing the effects of HBOT, apart from the mentioned psychological function tests, several ways of measuring the proposed molecular therapeutic effects come to mind. For instance, several biomarkers have been suggested, such as metalloproteases, VEGF, HIF1α, laminin-5, or interleukins. Moreover, a general heterogeneity and differences of regional cerebral oxygenation (rSO2) must be taken into account. Techniques such as near-infrared spectroscopy (NIRS) have in the past shown the ability to detect oxygenation responses of the brain during an after CA and CPR. It is not yet known whether NIRS can depict HBOT effects, but a hypothesis of "selective neuronal vulnerability" could be assessed through it. Lastly, endothelial dysfunction that has been reported to be occurring in CA patients, could be assessed via non-invasive function tests and biomarkers of endothelial function in order to depict the potential ameliorating effect of HBOT.

Knowledge gaps:

Lack of data on HBOT in immediate post ROSC patients: No randomized controlled study in humans has been carried out. There is an urgent need to determine the value of HBOT in the burden of CA and post CA pathologies. Insufficient data on HBOT in CA survivors: Preliminary data on HBOT in CA survivors are scarce, not robust, and highly heterogenic. Need for robust comparison data from healthy volunteers: Baseline values and potential normal dynamics of the outcome values must be acquired in individuals not being associated with CA to correctly interpret gained data from CA patients / survivors.

Experimental design Project aims: This is a pilot study that aims at general project feasibility. It should serve as a steppingstone for a large randomized controlled trial. Due to substantial costs and organizational efforts necessary for a larger trial, the pilot study is needed as a proof of concept beforehand. The goal of the overall project is to determine the effect of HBOT in a comprehensive approach towards resuscitation medicine, including comparison data from healthy volunteers. The pilot study should clarify feasibility (= primary outcome; defined as successfully recruiting the given number of individuals and successfully conducting the HBOT intervention) and potentially needed adaptations to the main study protocol in each study arm. The following main study will assess the primary null hypothesis "HBOT of any sub-kind is not associated with a beneficial dynamic in markers of inflammation" among assessing several other secondary outcomes (if deemed feasible in this pilot).

Secondary outcomes include the feasibility of integrating the HBOT study intervention into the ongoing clinical work, and successfully collecting further outcome values. These include (always obtained before and after treatment, except for the control groups): Baseline characteristics (all patients & probands; also including CA details); NIRS (ICU patients post ROSC, noninvasively) for assessing regional cerebral oxygen saturation and as a prognosticator after CA; PWV (all patients & probands, noninvasively): for assessing arterial stiffness at baseline and after a potential impact of the intervention as a marker of vessel remodeling and due to its link to inflammation and endothelial dysfunction; Laboratory markers (all patients and probands) for biobanking (35ml) including markers suggested by the study collaborators and past literature. Survival to hospital discharge and 30 days and 6 months; Neuropsychological testing; Neurological function; Health-related quality of life. All measured values eligible for follow-up are - in addition to the timepoint before HBOT - assessed again after HBOT.

Methodology: Randomized controlled pilot trial in a multiphase fashion. The study collective consists of three study arms: intensive care unit (ICU) patients after ROSC, healthy volunteers, and survivors of CA. ICU patients: Inclusion criteria: sustained ROSC since a maximum of 24 hours, hemodynamic and respiratory stable enough for transportation to HBOT. Exclusion criteria: traumatic CA, age <18 years, pregnancy, (tension-) pneumothorax. Healthy volunteers: Inclusion criteria: able to come to the study site themselves. Exclusion criteria: age <18 years, (suspected or desired) pregnancy, known chronic illnesses, especially known claustrophobia, history of CA, history of pneumothorax, acute or chronic ear / nose condition. CA survivors after hospital discharge: Inclusion criteria: history of CA from hospital discharge up to a maximum of 3 years ago, able to come to the study site themselves. Exclusion criteria: age <18 years, (suspected or desired) pregnancy, known claustrophobia, history of pneumothorax, acute or chronic ear / nose condition. Each study arm consists of three groups (one not receiving the intervention, one receiving HBOT only once, one receiving HBOT multiple times).

The intervention is defined as HBOT (carried out in the routine way that is well-established at the research facility). The details of the HBOT sessions with welcoming of the patient etc. cannot be described in detail in this short study overview.

Risks and Ethics: HBOT was repeatedly shown to provide antioxidant effects, balancing out the negative features. HBOT has therefore been described as safe due to its balance between oxidation and antioxidation. A safe practice of transporting the ICU patient to the hyperbaric chamber and monitoring them continuously during preparations and treatment itself is given at all times and provided by the ICU staff. Mechanical ventilation and various potentially necessary treatments of ICU patients have been decided to be feasible and safe in hyperbaric conditions, also by the European Committee for Hyperbaric Medicine. The desired pressure (2 ATM), has in the past been shown to be safe with a remarkably low incidence of side effects. Also, past research efforts have shown that the inclusion of healthy volunteers is both feasible and safe. A positive vote of the respective Ethics Committee of the research institution in Antwerp hqs already been obtained.

ELIGIBILITY:
Depending on the study arm.

ICU patients:

Inclusion criteria: sustained ROSC since a maximum of 24 hours, hemodynamic and respiratory stable enough for transportation to HBOT.

Exclusion criteria: traumatic CA, age <18 years, pregnancy, (tension-) pneumothorax.

Healthy volunteers:

Inclusion criteria: able to come to the study site themselves. Exclusion criteria: age <18 years, (suspected or desired) pregnancy, known chronic illnesses, especially known claustrophobia, history of CA, history of pneumothorax, acute or chronic ear / nose condition.

CA survivors after hospital discharge:

Inclusion criteria: history of CA from hospital discharge up to a maximum of 3 years ago, able to come to the study site themselves.

Exclusion criteria: age <18 years, (suspected or desired) pregnancy, known claustrophobia, history of pneumothorax, acute or chronic ear / nose condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study approach | 8 months
  Successfully recruiting at least 10 patients in each of the 3 study arms

SECONDARY OUTCOMES:
Inflammation dynamics | around 7 days (individual patient) / 8 months (study duration)
  interleukin-levels before- and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Koen Monsieurs, Prof., MD, Study Director — University Hospital of Antwerp, Belgium
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No